CLINICAL TRIAL: NCT05457257
Title: A Randomized, Open-label Study to Assess the Efficacy and Safety of Olaparib Versus Enzalutamide or Abiraterone Acetate in Chinese Men With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Prior Treatment With a New Hormonal Agent and Have BRCA1/2 Mutations (PROfound-CN)
Brief Title: Clinical Study to Assess the Efficacy and Safety of Olaparib in Chinese Patients With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Prior Treatment With a New Hormonal Agent and Have BRCA1/2 Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Foundation Medicine (Industry); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D081LC00002
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer (mCRPC); BRCA1/2 mutations
MeSH Terms: interventions — olaparib; enzalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olaparib (Experimental): Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Subjects will be administered study treatment orally at a dose of 300 mg twice daily (bid). The planned dose of 300 mg bid will be made up of two x 150 mg tablets twice daily, with 100 mg tablets used to manage dose reductions
  Interventions: Drug: olaparib
- Enzalutamide OR abiraterone acetate (Active Comparator): Enzalutamide:
  Enzalutamide is available as capsules or tablets containing 40 mg of enzalutamide. Subjects will be administered study treatment orally at a dose of 160 mg once daily.
  Abiraterone acetate with prednisone: Abiraterone acetate is available as tablets containing 250 mg of abiraterone acetate. Subjects will be administered study treatment orally at a dose of 1,000 mg once daily. Prednisone is 5mg twice daily. Prednisolone is permitted for use instead of prednisone if necessary.
  Interventions: Drug: enzalutamide; Drug: abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: olaparib — 300 mg (2x 150 mg tablets) twice daily
  Other Names: Lynparza
  Arms: Olaparib
Drug: enzalutamide — 160 mg (4 x 40 mg capsules) once daily
  Other Names: XTANDI
  Arms: Enzalutamide OR abiraterone acetate
Drug: abiraterone acetate — 1,000 mg (4 x 250 mg tablets) once daily
  Other Names: ZYTIGA
  Arms: Enzalutamide OR abiraterone acetate
Drug: Prednisone — 5mg(5mg x 1 tablet) twice daily
  Arms: Enzalutamide OR abiraterone acetate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Olaparib compared with standard of care (Enzalutamide or Abiraterone Acetate) in Chinese men with metastatic castration-resistant prostate cancer who have failed prior treatment with a new hormonal agent and have BRCA1/2 mutations.

DETAILED DESCRIPTION:
This is a Phase IV, randomized, open-label, 2-arm, multicenter study evaluating the efficacy and safety of olaparib in Chinese men with metastatic castration-resistant prostate cancer (mCRPC) who have failed prior treatment with a new hormonal agent (NHA) and have BRCA1/2 mutations. Approximately 42 subjects will be randomized in a 2:1 ratio to olaparib or to investigator's choice of NHA (enzalutamide or abiraterone acetate).

ELIGIBILITY:
Inclusion criteria：

1. Histologically confirmed diagnosis of prostate cancer.
2. Documented evidence of metastatic castration resistant prostate cancer (mCRPC).
3. Subjects must have progressed on prior new hormonal agent (e.g. abiraterone acetate and/or enzalutamide) for the treatment of metastatic prostate cancer and/or CRPC .
4. Ongoing therapy with LHRH analog or bilateral orchiectomy.
5. Radiological progression at study entry while on androgen deprivation therapy (or after bilateral orchiectomy).
6. Deleterious or suspected deleterious BRCA1/2 mutation in tumor tissue.
7. Normal organ and bone marrow function measured within 28 days prior to administration of study treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.

Exclusion criteria：

1. Any previous treatment with a poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor, including olaparib.
2. Subjects who had any previous treatment with DNA-damaging cytotoxic chemotherapy, except if for non-prostate cancer indication and last dose > 5 years prior to randomization.
3. History of another primary malignancy except for malignancy treated with curative intent with no known active disease for ≥5 years before the first dose of study intervention and of low potential risk for recurrence.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian Zhou, M.D., Principal Investigator — Sun Yat-sen University
Locations (28):
- China (28):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jiaxing
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wanzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment（https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure).
  "Yes" indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081LC00002&attachmentIdentifier=028f6e9b-9812-42c4-816e-2aa2bdf5c927&fileName=D081LC00002_-___Protocol_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081LC00002&attachmentIdentifier=8b69f6d0-0e93-4ef1-ac74-e8032da37880&fileName=D081LC00002_Profound_CN_SAP_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081LC00002&attachmentIdentifier=9f7fde03-5a07-4725-9eba-0b345f8cc650&fileName=d081lc00002-study-synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Olaparib 300 mg bd: Participants will receive olaparib 300 mg oral tablets, twice daily
- Investigators Choice of NHA: Participants will receive either enzalutamide 160 mg oral capsules/tablets once daily or abiraterone acetate 1000 mg oral tablets (plus prednisone 5 mg oral tablets twice daily)
Period: Overall Study
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Started | 29 | 14
Completed | 0 | 0
Not Completed | 29 | 14
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 10 | 3
Not completed — Ongoing | 19 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA | Total
Number analyzed (Participants) | 29 | 14 | 43
Age, Continuous [Median (Full Range); unit: Years] | 68.0 [56 to 82] | 67.5 [52 to 75] | 68.0 [52 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 14 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 14 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 29 | 14 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiological Progression-free Survival - Based on Blinded Independent Central Review (BICR)
Description: rPFS is defined as the time from randomization until the date of objective disease progression (soft tissue or bone) or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression.
Time Frame: Tumor assessments every 8 weeks (± 1 week) relative to the date of randomization until radiological progression as assessed by BICR or death (median duration of treatment of 9 and 6 months for Olaparib and Investigators Choice of NHA respectively).
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Months | 9.331 [5.65 to 11.20] | 8.838 [1.77 to NA] — NA - not calculated as an insufficient number of events for the upper limits of the 95% confidence interval
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Investigators Choice of NHA; The explanation of statistical method; Test type: Superiority; p = 0.726, Log Rank — The 2-sided nominal p-values were calculated using the log-rank test stratified by the same variables selected in the primary pooling strategy, using the Breslow method for handling ties; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.46 to 3.45] — The Hazard ratio and CI were calculated using a Cox Proportional Hazards model adjusted for the variables. The Efron approach was used for handling ties. A hazard ratio <1 favours Olaparib 300 mg bd

2. Secondary Outcome: Confirmed Objective Response Rate (ORR), Based on Blinded Independent Review (BICR)
Description: Confirmed ORR is the percentage of patients with a Complete response (CR) or Partial response (PR), in their soft tissue disease per (RECIST v1.1), in the absence of progression on bone scan per Prostate Cancer Working Group 3 (PCWG3), confirmed >=4 weeks later. Per RECIST v1.1, CR=Disappearance of all target lesions; PR = >=30% decrease in the sum of diameters of target lesions. For each treatment group, confirmed ORR is the number of patients with a confirmed CR or PR divided by the number of patients in the treatment group.
Time Frame: Tumor assessments every 8 weeks (± 1 week) from randomisation until radiographic progression assessed by BICR (median duration of treatment of 9 and 6 months for Olaparib and Investigators Choice of NHA respectively).
Population: Evaluable for response analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 12 | 5
Participants | 5 | 1
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Investigators Choice of NHA; The explanation of statistical method; Test type: Superiority; p = 0.498, Regression, Logistic — A Fisher's exact test using mid p-values was used; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.20 to 59.66] — Objective response rate compared using logistic regression adjusting for previous taxane use as a covariate. An odds ratio >1 favours Olaparib 300 mg bd. CI calculated using profile likelihood method

3. Secondary Outcome: Overall Survival
Description: OS is the time from the date of randomization until death due to any cause.
Time Frame: From the time from the date of randomization until death due to any cause. Assessments continue up to 27 months after the first patient was randomized.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Months | 17.314 [13.90 to NA] — NA - not calculated as an insufficient number of events for the upper limits of the 95% confidence interval | NA [10.32 to NA] — NA - Not calculated, estimate cannot be calculated as the median OS was not reached. Insufficient number of participants with events for median and upper limits of 95% confidence interval.
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Investigators Choice of NHA; The explanation of statistical method; Test type: Superiority; p = 0.440, Log Rank — The 2-sided nominal p-values were calculated using the log-rank test stratified by the same covariates and using the Breslow method for handling ties; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.50 to 7.48] — The hazard ratio and CI were calculated using a Cox Proportional Hazards model with the Efron approach being used for handling ties, adjusting for covariates. A hazard ratio <1 favours Olaparib 300 mg bd

4. Secondary Outcome: Time to First Symptomatic Skeletal-related Event
Description: Time from first dose to the first symptomatic skeletal-related event
Time Frame: Time from randomization to the first SSRE-radiation for skeletal symptoms, confirmed pathological fracture, confirmed spinal cord compression, or orthopaedic surgery for bone metastases. Assessments continue up to 27 months post first patient enrolled.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Months | NA [NA to NA] — NA - Not calculated, estimate cannot be calculated as the median SSRE was not reached. Insufficient number of participants with events for median and lower and upper limits of 95% confidence interval. | NA [NA to NA] — NA - Not calculated, estimate cannot be calculated as the median SSRE was not reached. Insufficient number of participants with events for median and lower and upper limits of 95% confidence interval.

5. Secondary Outcome: Time to Opiate Use for Cancer-related Pain
Description: Time from randomization to opiate use for cancer-related pain
Time Frame: Opioid use will be recorded at baseline and at every study visit, including the safety follow-up visit. Assessments continue up to 27 months post first patient enrolled.
Population: Full analysis set (Only includes patients who were not on opiates at baseline)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 23 | 9
Months | NA [11.20 to NA] — NA - Not calculated, estimate cannot be calculated as the median Opioid use free was not reached. Insufficient number of participants with Opioid use free for median and upper limits of 95% confidence interval. | 17.281 [1.31 to NA] — NA - Not calculated as an insufficient number of participants with Opioid use free for upper limits of 95% confidence interval.
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Investigators Choice of NHA; The explanation of statistical method; Test type: Superiority; p = 0.604, Log Rank — The 2-sided nominal p-value was calculated using the log-rank test stratified by the same variables selected in the primary pooling strategy, using the Breslow method for handling ties; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.20 to 2.88] — The Hazard ratio and CI were calculated using a Cox Proportional Hazards model adjusted for the variables selected in the primary pooling strategy: none. The Efron approach was used for handling ties. A hazard ratio <1 favours Olaparib 300 mg bd

6. Secondary Outcome: Prostate-specific Antigen Response
Description: Proportion of participants achieving a ≥50% decrease in PSA from baseline to the lowest post-baseline PSA result, confirmed by a second consecutive PSA assessment at least 3 weeks later (PSA50 response)
Time Frame: Blood samples for PSA assessment will be collected at baseline and every 4 weeks throughout the treatment phase, including at the study treatment discontinuation visit. Assessments continue up to 27 months post first patient enrolled.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Percentage of participants
  Single visit response | 48 [29 to 67] | 36 [13 to 65]
  Confirmed response | 41 [24 to 61] | 29 [8 to 58]

7. Secondary Outcome: Prostate-specific Antigen Response
Description: Best percentage change from baseline in PSA is defined as the biggest reduction in PSA level compared with baseline (or the smallest increase in the absence of a reduction) taking account of all PSA values collected for each patient.
Time Frame: as for outcome 6
Population: Full Analysis Set (Only includes patients have baseline PSA and post-baseline PSA results for analysis of "Best percentage change from baseline" and includes patients have baseline PSA and week 12 PSA for analysis of "Percentage change from baseline at Week 12" )
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Percentage change from baseline
  Percentage change from baseline at Week 12: number analyzed (Participants) | 22 | 7
  Percentage change from baseline at Week 12 | 37.2 (252.62) | -15.0 (53.84)
  Best percentage change from baseline: number analyzed (Participants) | 26 | 12
  Best percentage change from baseline | -40.6 (60.06) | -22.7 (74.62)

8. Secondary Outcome: Time From Randomization to Second Progression or Death
Description: Time from randomization to second progression by investigator assessment of radiological or clinical progression or death (PFS2)
Time Frame: Tumor assessments will be performed every 8 weeks (±7 days) after randomization until radiologic progression or death, unless the participant withdraws consent. Assessments continue up to 27 months post first patient enrolled.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Months | NA [15.41 to NA] — NA - Not calculated, estimate cannot be calculated as the median PFS2 was not reached. Insufficient number of participants with events for median and upper limits of 95% confidence interval. | NA [5.91 to NA] — NA - Not calculated, estimate cannot be calculated as the median PFS2 was not reached. Insufficient number of participants with events for median and upper limits of 95% confidence interval.
Statistical Analysis 1: Comparison: Olaparib 300 mg bd vs Investigators Choice of NHA; The explanation of statistical method; Test type: Superiority; p = 0.889, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.19 to 6.24] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Subsequent Anticancer Therapy
Time Frame: Recorded from post discontinuation of study treatment up to primary data cut off date. Assessments continue up to 27 months post first patient enrolled.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd | Investigators Choice of NHA
Number analyzed (Participants) | 29 | 14
Participants
  Any post-discontinuation anti-cancer therapy | 14 | 3
  Immunotherapy | 0 | 0
  Hormonal therapy | 12 | 2
  Taxane chemotherapy | 4 | 0
  Platinum chemotherapy | 0 | 0
  PARP inhibitor | 0 | 3
  Other | 1 | 0

ADVERSE EVENTS:
Time Frame: From the time of signature of the ICF, throughout the treatment period and until the 30-day follow-up period is completed or 27 months post first patient enrolled, whichever occurs earlier
Groups:
- Olaparib 300mg bd: Description (Arm-group)
Arm/Group | Olaparib 300mg bd | Investigators Choice of NHA
All-Cause Mortality (participants affected / at risk) | 10/29 | 3/14
Serious Adverse Events (participants affected / at risk) | 13/29 | 5/14
Other Adverse Events (participants affected / at risk) | 28/29 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg bd (N=29) | Investigators Choice of NHA (N=14)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg bd (N=29) | Investigators Choice of NHA (N=14)
Constipation (Gastrointestinal disorders) | 7 (8) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (10) | 4 (4)
Asthenia (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 22 (23) | 5 (5)
Malaise (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Bilirubin excretion disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Adenosine deaminase increased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Blood creatinine increased (Investigations) | 4 (5) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 2 (3)
Eastern cooperative oncology group performance status worsened (Investigations) | 2 (2) | 0 (0)
Eosinophil count decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (13) | 2 (2)
Neutrophil count decreased (Investigations) | 6 (14) | 3 (7)
Platelet count decreased (Investigations) | 6 (9) | 3 (5)
Urinary occult blood positive (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 7 (7) | 3 (4)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 7 (15) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (6) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (10) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT05457257/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT05457257/SAP_001.pdf